CLINICAL TRIAL: NCT00877669
Title: The Comparison of Efficacy Between Holmium Laser Enucleation of the Prostate (HoLEP) and Transurethral Resection of the Prostate (TURP) on the Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostate Hyperplasia (BPH)
Brief Title: Efficacy Study of HoLEP and TURP on LUTS Secondary to BPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Urology, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-10-038
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transurethral resection of the prostate (Active Comparator): TURP group
  Interventions: Procedure: Transurethral resection of the prostate
- Holmium Laser Enucleation of Prostate (Experimental): HoLEP group
  Interventions: Procedure: Holmium Laser Enucleation of the Prostate

INTERVENTIONS:
Procedure: Transurethral resection of the prostate — Standard transurethral resection of the prostate using electrocautery loop
  Other Names: TURP
  Arms: Transurethral resection of the prostate
Procedure: Holmium Laser Enucleation of the Prostate — HoLEP using 100W Ho:YAG laser
  Arms: Holmium Laser Enucleation of Prostate

SUMMARY:
The purpose of this study is to compare of Efficacy and Safety Between Holmium Laser Enucleation of the Prostate (HoLEP) and Transurethral Resection of the Prostate (TURP) on the Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostate Hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* 50 yrs or greater
* International prostatic symptom score >= 12
* Bladder outlet obstruction confirmed by pressure-flow study (BOOI > 20)
* Able to give fully informed consent

Exclusion Criteria:

* Patients with urologic malignancies such as prostate cancer and bladder cancer
* Patients underwent urethral, prostate surgery
* Patients with urethral stricture or bladder diverticulum or bladder neck contracture
* Patients with histories of bacterial prostatitis within 1 year
* seems not to be appropriate to this study by the decision of investigators because of any other reasons

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2008-10; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The changes of International Prostatic Symptom Scores (IPSS) from baseline to 6 months after operation | 6 months

SECONDARY OUTCOMES:
The changes of Quality of Life (QoL) parameters | 6 months
The changes of IPSS and QoL parameters | 1 month and 3months after operation
The changes of Uroflowmetry (UFM) and Postvoid residual urine(PVR) parameters | 2 weeks and 3 and 6 months after operation
Postoperative hospital stay days and postoperative catheterization days | immediate postoperative period
The changes of the hemoglobin and the serum sodium | 0 and 1 day after operation
Operative time and Resected tissue weight | 0 day after operation
The changes of ICS male questionnaire (short form) parameters | 3 and 6 months after operation
The changes of international index of erectile function (IIEF)-15 parameters | 6 months after operation
The changes of Patient perception of treatment benefit questionnaire (PPTB) parameters | 3 and 6 months after operation
The changes of voiding frequencies and urgency parameters in Frequency volume chart | 3 and 6 months after operation
Ejaculation parameter | 6 months after operation
Complications | During all study periods

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D.,M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea